CLINICAL TRIAL: NCT03614039
Title: Effect of Alive Probiotics Supplementation With Absorbent Smectite Gel in NAFLD
Brief Title: Effect of Probiotic and Smectite Gel on NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarii Kobyliak (Other)
Responsible Party: Sponsor-Investigator, Nazarii Kobyliak, Associate Professor of Endocrinology Department, PhD, Bogomolets National Medical University
Organization: Bogomolets National Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-3
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases; Digestive System Diseases; Type2 Diabetes
Keywords: diosmectite; nutraceuticals; non-alcoholic fatty liver disease; probiotics; Lactobacillus; Bifidobacterium; Propionibacterium
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases; Digestive System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic-smectite (Active Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day.
  Interventions: Dietary Supplement: "Symbiter Forte"
- placebo (Placebo Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: "Symbiter Forte" — "Symbiter Forte" which contains combination of smectite gel (250 mg), and biomass of 14 alive probiotic strains: Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g)
  Arms: probiotic-smectite
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
Smectite is a natural silicate clay belonging to the dioctahedral smectite class and has the ability directly to absorb bacterial toxins, bacteria, viruses and bile salts. Diosmectite also has a protective effect against intestinal inflammation hence suppressing production of cytokines such as IL-8 and TNFα. Investigators suggested that all these pharmacological properties may be beneficial for the treatment of NAFLD. Based on preclinical data, in rats with MSG induced obesity supplementation of alive probiotics with smectite gel (Symbiter-Forte) due to his absorbent activity lead to significant reduction of chronic systemic inflammatory markers, lower total NAS (NAFLD activity score) score, with more pronounced reduction of lobular inflammation as compared to administration of probiotic alone. In respect to preclinical data, in this double-blind single center randomized clinical trial (RCT) the efficacy of alive probiotics supplementation with smectite gel (Symbiter-Forte) vs. placebo in type-2 diabetes patient with NAFLD detected on ultrasonography will be studied

DETAILED DESCRIPTION:
In this single-center double-blind, placebo controlled, parallel group study, 50 T2D patients from the Kyiv City Clinical Endocrinology Center - Ukraine, were selected. They were randomly assigned to receive "Symbiter Forte" or placebo for 8 weeks, administered as a sachet formulation in double-blind treatment. Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.

The "Symbiter Forte" was supplied by Scientific and Production Company "O.D. Prolisok". It contains combination of smectite gel (250 mg), supplemented with biomass of 14 alive probiotic strains: Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patients received 1 sachet (10 grams) of probiotic-smectite and placebo per day. All sachets were identical with similar organoleptic characteristics (e.g., taste and appearance).

The pre-randomization period was designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study started, after the informed consent was signed, patients were instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants were instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent the study were instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits were provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy was compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-75, BMI ≥25 kg/m2) diagnosed with NAFLD according to the recommendations of the American Gastroenterology Association (AGA) and American Association for the Study of Liver Disease (AASLD);
* the diagnosis of fatty liver was based on the results of abdominal ultrasonography. Of 4 known criteria (hepato-renal echo contrast, liver brightness, deep attenuation, and vascular blurring), the participants were required to have hepato-renal contrast and liver brightness to be given a diagnosis of NAFLD.
* type 2 diabetes treated with diet and exercise alone or metformin, SUs and insulin at stable dose at least 4 weeks prior to the commencement of the study;
* AST and ALT ≤3x upper limit of normal.

Exclusion Criteria:

* alcohol abuse (>20 g/day (2 standard drinks) in women or > 30 g/d (3 drinks) in men over a two-year period);
* chronic viral hepatitis (associated with HBV, HCV, HDV infection);
* drug-induced liver disease, Wilson's disease, hereditary deficiency of antitrypsin-1 and idiopathic hemochromatosis;
* history of decompensated liver disease including ascites, encephalopathy or variceal bleeding;
* regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment;
* antibiotic use within 3 months prior to enrollment;
* uncontrolled cardiovascular or respiratory disease, active malignancy, or chronic infections;
* use of agents such as vitamin E, omega-3 fatty acids or medications with evidence for effects on NAFLD (pioglitazone, GLP-1 analogues, dipeptidyl peptidase IV inhibitors, ursodeoxycholic acid);
* presence of active infection, pregnancy or lactation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
fatty liver index (FLI) | 8 weeks compared to baseline
  FLI = [e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745) / (1 + e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745)] × 100
liver stiffness (LS) | 8 weeks compared to baseline
  liver stiffness (LS) was measured by Shear Wave Elastography (SWE) and expressed in kPa

SECONDARY OUTCOMES:
ALT | 8 weeks compared to baseline
  ALT in IU/L
AST | 8 weeks compared to baseline
  AST in IU/L
γ-GT | 8 weeks compared to baseline
  γ-GT in IU/L
Total Cholesterol (TC) | 8 weeks compared to baseline
  TC in mmol/l
Tryglicerides (TG) | 8 weeks compared to baseline
  TG in mmol/l
LDL-Cholesterol (LDL-C) | 8 weeks compared to baseline
  LDL-C in mmol/l
VLDL-Cholesterol (VLDL-C) | 8 weeks compared to baseline
  VLDL-C in mmol/l
HDL-Cholesterol (HDL-C) | 8 weeks compared to baseline
  HDL-C in mmol/l
cytokines levels | 8 weeks compared to baseline
  TNF-α, IL-1β, IL-6, IL-8, INF-γ in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Petro Bodnar, Prof, Principal Investigator — Bogomolets National Medical University

IPD SHARING:
Plan to Share IPD: No